CLINICAL TRIAL: NCT05714917
Title: Longitudinal Assessment of Neurological Recovery in Patients Following Nitrous Oxide Abuse
Brief Title: Neurological Recovery Following NOS-SACD
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Barts & The London NHS Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22NS021
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Nitrous Oxide Abuse; Subacute Combined Cord Degeneration; Neurologic Symptoms; Paresthesia; B12 Deficiency Vitamin
Keywords: Nitrous oxide; B12; Neurological symptoms; Clinical recovery
MeSH Terms: conditions — Neurologic Manifestations; Paresthesia; Vitamin B 12 Deficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Confirmed diagnosis of NOS-induced neurological damage: Any patient first presented with paraesthesia, weakness, ataxia or gait disturbance with a history of NOS use (age limit 16-40) as of 19/08/2024.
  Patients who can read and write in English, so that they can complete the questionnaires.
  Interventions: Other: Observational study with no interventions

INTERVENTIONS:
Other: Observational study with no interventions — This is an observational study and there will be no clinical interventions.
  Other Names: Observational Study

SUMMARY:
Nitrous oxide has become an increasingly popular recreational drug amongst young people, particularly at festivals, nightclubs and parties. Considering the drug is not illegal to possess, has low cost in the form of 'whippets' and can be easily purchased online, it has become the second most commonly used recreational drug amongst people aged 16-24 in the UK. However, nitrous oxide is known to irreversibly inactivate the functioning of vitamin B12, a vitamin required for the maintenance and proper functioning of nerves in the spinal cord. Neurological symptoms in this population have been reported in around 3.4% of nitrous oxide users, although the true incidence is expected to be higher as the cases being reported by UK hospitals continues to rise.

Patients may present with adverse neurological symptoms like tingling, weakness, coordination and mobility problems. Currently, studies reviewing the functional recovery of these patients have been limited by a retrospective study design, short follow up duration and being limited to small cohort sizes. This is in part linked to patient non-compliance and non-attendance at follow-up appointments. The investigators will therefore prospectively recruit all patients presenting with these symptoms and continue to collect data relating to their neurological recovery for 12 months. Data collection will be remote to ensure it is of low burden to the participants. This will allow the investigating team and others to fully appraise the severity of these toxic neuropathies and understand how best to manage their follow up.

DETAILED DESCRIPTION:
This study will take place in selected participating hospitals, including their acute neurology units and emergency departments. Participants presenting to their GP will be referred per standard clinical care with the acute neurology units for study inclusion review. Ideally in all cases the investigating team would prefer for participants to be in hospitals (either directly through A&E or being referred by their GP to the acute neurology service) at the time of study inclusion and for the baseline visit to ensure standard clinical care data can be collected (including MRI, bloods and treatment information including how many Vitamin B12 injections are given at admission and throughout their recovery). Care will be taken over by the neurology team where possible and standard clinical practice for participants with NOS induced neurological damage will be managed and treated as per their own local guidelines. Patients identified to the research team with consultant confirmed NOS-induced neuropathy but have left hospital can still be considered for the study but oral consent will be asked of these participants.

Baseline visit: participants who remain in hospital at the time of study invite will have their concomitant medications, comorbidities and a neurological assessment reviewed in person, blood and MRI results will also be collected from the routine tests that have been performed whilst in hospital. Participants not in the hospital at this point will have this information assessed where possible via the telephone or obtained from their medical records. Individuals without blood or MRI data will not be excluded from the study providing they meet the inclusion criteria.

At the point of consent (written or verbal), recruited participants details (NHS number, name and mobile number) will be securely shared with the coordinating Nottingham University Hospitals NHS Trust center. The Nottingham researcher will then add new participants to the PsychoPy platform which is the University of Nottingham spinoff company that allows remote clinical trial assessments. Each time a participant is added, the platform will automatically generate follow up dates for when each of the subsequent visits are due (baseline visit, 1-month, 3- month, 6-month and 12-month). The Nottingham coordinating team will generate a specific link from this platform each time a participant visit is due, the link will then be sent via text messaging from the coordinating centre to the participants mobile phone. These links can be opened and the visits completed from anywhere provided the participant has internet connection. The content of the visits will include: demographic [baseline visit only], NOS quantification, basic finger tapping task, cognitive function tasks, health questionnaire assessing participants ability to perform simple daily activities, the overall neuropathy limitations scale and the average step count for the last 7-days.

The coordinating team will continue to monitor completed and outstanding visits for all participants and where uncompleted, will send out reminder text messages to the participants.

Our pragmatic approach to perform only remote follow ups was based on the already previously reported high DNA rate in this patient population. All patients will participate in a total of 5 remote visit assessments over the 12-month period.

A nested qualitative sub-study is being led by Professor Alastair Noyce and Dr Laura Smith, based at Queen Mary University of London. Semi-structured interviews will be undertaken with participants taking part in the longitudinal cohort study, who have agreed to be contacted about allied research opportunities. Interviews will cover their lived experiences of using NOS, any mental health difficulties experienced, and explore any links between these two areas. Participants will also be asked about any treatment accessed for NOS usage and mental health difficulties, and explore the barriers and facilitators to engagement with treatment. We will collect qualitative data at any point after the participant has provided informed consent for the qualitative sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient first presented with paraesthesia, weakness, ataxia or gait disturbance with a history of NOS use (age limit 16-40) as of 19/08/2024
* Patients who can read and write in English, so that they can complete the questionnaires.
* Patients must have received a definitive consultant neurologist confirmed diagnosis of NOS-induced neurological damage. This is possible as all eligible patients will have been reviewed by the neurology team prior to study involvement.

Exclusion Criteria:

•Other causes of previous neuropathy or neurodegeneration indicated.

Qualitative Interview Study:

* Patients currently taking part in the longitudinal study.
* Patients who report previously (clinical history) or currently (PHQ-2, clinical history) experiencing mental health difficulties.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: NOS induced neurological symptoms may present with either a.) severe neurological impairment to warrant A&E admission, or b.) milder symptoms which may present to primary care. The investigators team therefore propose recruitment pathways based either on A&E or GP referral. Participants will be invited to the neurology team in order for them to coordinate the care according to local practices.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Improvement in finger tapping task, baseline to month 12 | 12 months
  To determine whether patients with NOS-induced neurological damage recover their dexterity function over a 12-month period.

SECONDARY OUTCOMES:
Improvement in cognitive function task, baseline to month 12 | 12 months
  To determine whether patients with NOS-induced neurological damage recover their cognitive function over a 12-month period.
Improvement in step counts, baseline to month 12 | 12 months
  To determine whether patients with NOS-induced neurological damage recover their average weekly step counts over a 12-month period.
Improvement in I-RODS and ONLS, baseline to month 12 | 12 months
  To determine whether patients with NOS-induced neurological damage recover their neuropathy and general health scores over a 12-month period.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health NHS Trust, London
  - Salford Royal NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
The study team have not yet established a plan to share IPD.

REFERENCES:
- [Background] Kroes AC, Lindemans J, Abels J. [Interaction between nitrous oxide and vitamin B12]. Ned Tijdschr Geneeskd. 1985 Nov 23;129(47):2243-7. No abstract available. Dutch. PMID 4088327
- [Background] Omotosho YB, Ying GW, Orji R, Patel H. Recreational Nitrous Oxide-Induced Subacute Combined Degeneration. Cureus. 2022 Mar 22;14(3):e23409. doi: 10.7759/cureus.23409. eCollection 2022 Mar. PMID 35475085
- [Background] Winstock AR, Ferris JA. Nitrous oxide causes peripheral neuropathy in a dose dependent manner among recreational users. J Psychopharmacol. 2020 Feb;34(2):229-236. doi: 10.1177/0269881119882532. Epub 2019 Nov 4. PMID 31679459
- [Background] Schilling RF. Is nitrous oxide a dangerous anesthetic for vitamin B12-deficient subjects? JAMA. 1986 Mar 28;255(12):1605-6. PMID 3951096
- [Background] Flippo TS, Holder WD Jr. Neurologic degeneration associated with nitrous oxide anesthesia in patients with vitamin B12 deficiency. Arch Surg. 1993 Dec;128(12):1391-5. doi: 10.1001/archsurg.1993.01420240099018. PMID 8250714
- [Background] Patel KK, Mejia Munne JC, Gunness VRN, Hersey D, Alshafai N, Sciubba D, Nasser R, Gimbel D, Cheng J, Nouri A. Subacute combined degeneration of the spinal cord following nitrous oxide anesthesia: A systematic review of cases. Clin Neurol Neurosurg. 2018 Oct;173:163-168. doi: 10.1016/j.clineuro.2018.08.016. Epub 2018 Aug 9. PMID 30144777
- [Background] Seed A, Jogia M. Lessons of the month: Nitrous oxide-induced functional vitamin B12 deficiency causing subacute combined degeneration of the spinal cord. Clin Med (Lond). 2020 May;20(3):e7-e9. doi: 10.7861/clinmed.2020-0072. PMID 32414730
- [Background] de Medeiros FC, de Albuquerque LA, de Souza RB, Gomes Neto AP, Christo PP. Vitamin B12 extensive thoracic myelopathy: clinical, radiological and prognostic aspects. Two cases report and literature review. Neurol Sci. 2013 Oct;34(10):1857-60. doi: 10.1007/s10072-013-1335-7. Epub 2013 Mar 7. PMID 23468407
- [Background] Algahtani H, Shirah B, Abdelghaffar N, Abuhawi O, Alqahtani A. Nitrous oxide recreational abuse presenting with myeloneuropathy and mimicking Guillain-Barre syndrome. Intractable Rare Dis Res. 2020 Feb;9(1):54-57. doi: 10.5582/irdr.2020.01007. PMID 32201677
- [Background] Swart G, Blair C, Lu Z, Yogendran S, Offord J, Sutherland E, Barnes S, Palavra N, Cremer P, Bolitho S, Michael Halmagyi G. Nitrous oxide-induced myeloneuropathy. Eur J Neurol. 2021 Dec;28(12):3938-3944. doi: 10.1111/ene.15077. Epub 2021 Sep 6. PMID 34427020
- [Background] Berling E, Fargeot G, Aure K, Tran TH, Kubis N, Lozeron P, Zanin A. Nitrous oxide-induced predominantly motor neuropathies: a follow-up study. J Neurol. 2022 May;269(5):2720-2726. doi: 10.1007/s00415-021-10858-2. Epub 2021 Nov 6. PMID 34741241
- [Background] Garakani A, Jaffe RJ, Savla D, Welch AK, Protin CA, Bryson EO, McDowell DM. Neurologic, psychiatric, and other medical manifestations of nitrous oxide abuse: A systematic review of the case literature. Am J Addict. 2016 Aug;25(5):358-69. doi: 10.1111/ajad.12372. Epub 2016 Apr 1. PMID 27037733
- [Background] Zheng D, Ba F, Bi G, Guo Y, Gao Y, Li W. The sharp rise of neurological disorders associated with recreational nitrous oxide use in China: a single-center experience and a brief review of Chinese literature. J Neurol. 2020 Feb;267(2):422-429. doi: 10.1007/s00415-019-09600-w. Epub 2019 Oct 26. PMID 31655888
- [Background] Peirce J, Gray JR, Simpson S, MacAskill M, Hochenberger R, Sogo H, Kastman E, Lindelov JK. PsychoPy2: Experiments in behavior made easy. Behav Res Methods. 2019 Feb;51(1):195-203. doi: 10.3758/s13428-018-01193-y. PMID 30734206
- See also: Drug misuse in England and Wales - Office for National Statistics — https://www.ons.gov.uk/peoplepopulationandcommunity/crimeandjustice/articles/drugmisuseinenglandandwales/yearendingmarch2020#trends-in-use-of-individual-drug-types
- See also: Global Drug Survey 2021 — https://www.globaldrugsurvey.com/wp-content/uploads/2021/12/Report2021_ExecutiveSummary.pdf